CLINICAL TRIAL: NCT02653365
Title: Predictors of Non-invasive Ventilation Failure in Patients With Acute Cardiogenic Pulmonary Edema
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zujin Luo, Attending physician, Beijing Chao Yang Hospital
Other Study IDs: BeijingCYH-ICU-002
Record Dates: First submitted 2015-12-24; First posted 2016-01-12 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Acute Cardiogenic Pulmonary Edema
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Non-invasive ventilation: All patients eligible for inclusion in the study were treated with Non-invasive ventilation.
  Interventions: Device: Non-invasive ventilation

INTERVENTIONS:
Device: Non-invasive ventilation — Noninvasive ventilation (NIV) was performed with a noninvasive ventilator (BiPAP Synchrony®, Respironics Inc., Murrysville, PA, USA).

SUMMARY:
The aims of our study was to identify early predictors of non-invasive ventilation failure, so as to alert clinicians early that endotracheal intubation and mechanical ventilation might be appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ACPE diagnosed based on SpO2 below 90% with >5 L/ min oxygen via reservoir face mask
* Acute respiratory distress as evidenced by severe dyspnea
* Breathing frequency of >30 breaths/min, and use of accessory respiratory muscles or paradoxical abdominal motion in association with tachycardia
* Cardiac gallops, bilateral rales, and typical findings of congestion on chest radiography, without a history suggesting pulmonary aspiration or evidence of pneumonia.

Exclusion Criteria:

* Patients were excluded from the study if they were intubated before ICU admission, or required immediate intubation without prior NIV, or presented a respiratory or cardiac arrest
* Severe hemodynamic instability (systolic arterial pressure <70 mmHg despite adequate fluid repletion and use of vasoactive agents) or life-threatening ventricular arrhythmias.
* Patients were also excluded if they were unresponsive, agitated, and unable to cooperate; or if they had any condition that precluded application of a face mask including upper airway obstruction
* Recent oral or facial trauma or surgery
* Recent gastric or esophageal surgery
* Inability to clear respiratory secretions or high risk for aspiration.
* In addition, patients were excluded if they had a "do not intubate" order or refused research authorization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ACPE
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Age | From study entry to death or intensive care unit (ICU) discharge, up to 3 years.
Heart rate | From study entry to death or ICU discharge, up to 3 years.
Blood pressure | From study entry to death or ICU discharge, up to 3 years.
Breath frequency | From study entry to death or ICU discharge, up to 3 years.
Arterial blood gas | From study entry to death or ICU discharge, up to 3 years.
New York Heart Association classification | From study entry to death or ICU discharge, up to 3 years.
  The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure.
  Class I: Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. no shortness of breath when walking, climbing stairs etc.
  Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Killip classification | From study entry to death or ICU discharge, up to 3 years.
  The Killip classification is a system used in individuals with an acute myocardial infarction, in order to risk stratify them. Patients were ranked by Killip class in the following way:
  Killip class I includes individuals with no clinical signs of heart failure. Killip class II includes individuals with rales or crackles in the lungs, an S3, and elevated jugular venous pressure.
  Killip class III describes individuals with frank acute pulmonary edema. Killip class IV describes individuals in cardiogenic shock or hypotension (measured as systolic blood pressure lower than 90 mmHg), and evidence of peripheral vasoconstriction (oliguria, cyanosis or sweating).
Left ventricular ejection fraction | From study entry to death or ICU discharge, up to 3 years.
B-type natriuretic peptide | From study entry to death or ICU discharge, up to 3 years.
Fluid balance within 24 hours after presence of acute cardiogenic pulmonary edema. | From study entry to death or ICU discharge, up to 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Institute of Respiratory Medicine, Department of respiratory and critical care medicine, Beijing Chao-Yang Hospital Jingxi Campus, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Luo Z, Han F, Li Y, He H, Yang G, Mi Y, Ma Y, Cao Z. Risk factors for noninvasive ventilation failure in patients with acute cardiogenic pulmonary edema: A prospective, observational cohort study. J Crit Care. 2017 Jun;39:238-247. doi: 10.1016/j.jcrc.2017.01.001. Epub 2017 Jan 6. PMID 28110770